CLINICAL TRIAL: NCT00872144
Title: A Double Blind Placebo Controlled Crossover Pilot Trial of Sativex With Open Label Extension for Treatment of Chemotherapy Induced Neuropathic Pain
Brief Title: Sativex for Treatment of Chemotherapy Induced Neuropathic Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mary Lynch (Other)
Responsible Party: Sponsor-Investigator, Mary Lynch, MD FRCPC, Nova Scotia Health Authority
Organization: Nova Scotia Health Authority (Other)
Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CDHA-RS/2009-316
Record Dates: First submitted 2009-03-25; First posted 2009-03-31 (Estimated); Last update posted 2014-03-07 (Estimated); Status verified 2014-03

CONDITIONS: Neuropathic Pain
MeSH Terms: conditions — Neuralgia | interventions — nabiximols

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sativex (Active Comparator)
  Interventions: Drug: Sativex

INTERVENTIONS:
Drug: Sativex — Sativex (or placebo) will be dispensed identical 5.5 ml containers. Participants will be instructed to start with a dose of 1 spray trans-mucosally at 1800 hrs. If there are no limiting adverse effects such as sedation or dizziness, participants will be instructed to increase the dose to 2 sprays- one in the morning and the other in the early evening on day two. Participants may increase the dose by 1-2 sprays per day to a maximum dose of 12 sprays per day given 3 sprays 4 times per day. In the initial titration phase participants will be instructed to space each dose actuation 15 minutes apart until accustomed to the preparation. Participants will titrate the dose to a level where they obtain an analgesic effect without limiting side effects.

SUMMARY:
Chemotherapy is often used to treat cancer and in many cases can cure it or extend life. Unfortunately many of the chemotherapeutic agents used in treating cancer can cause nerve damage, resulting in severe pain involving the extremities. This "neuropathic" pain causes significant suffering in cancer survivors and may also limit the amount of chemotherapy patients are able to tolerate in attempting to treat the cancer. There is evidence that cannabinoids can suppress chemotherapy evoked neuropathy in animal models, in some cases better than morphine. This study proposes to examine the effect of a cannabinoid extract (Sativex) in treatment of neuropathic pain caused by chemotherapy.

DETAILED DESCRIPTION:
The problem of neuropathic pain:

A recent review has identified a neuropathic pain prevalence rate of 2-3% in the general population 1. Based on a Canadian population of 30 million, this means that close to one million Canadians suffer with neuropathic pain. Neuropathic pain is one of the most difficult types of persistent pain to treat effectively. No more than 50% 2 of patients with neuropathic pain obtain adequate relief using current treatments. This is related to the fact that there are numerous pathophysiological mechanisms that contribute to neuropathic pain. Neuropathic pain is now understood to involve neural responses in which both peripheral and central mechanisms contribute to the generation of spontaneous pain and evoked aspects including allodynia and hyperalgesia 3-5, Traditional approaches to neuropathic pain have involved the use of oral medications as single agents or in combination (NSAIDs, opioids, anticonvulsants, tricyclic type antidepressants) 6,7. Unfortunately this approach is often inadequate and accompanied by side effects. New treatments are needed for management of neuropathic pain

Neuropathic pain associated with chemotherapy:

Neuropathic pain associated with chemotherapy used for treatment of solid tumors (eg. paclitaxil, vincristine and cis-platin) is particularly resistant to treatment and is a growing clinical problem as chemotherapeutic regimes grow more successful in extending life. This type of neuropathic pain is particularly resistant to treatment and contributes to the overall level of suffering experienced by patients who recovering from cancer treatment with chemotherapy. There is pre-clinical evidence supporting that cannabinoid agonists may be helpful for treatment neuropathic pain caused by chemotherapy.

Cannabinoids in treatment of pain:

The potent anti-nociceptive and antihyperalgesic effects of cannabinoid agonists in animal models of acute and chronic pain, the presence of cannabinoid receptors in pain-processing areas of the brain, spinal cord and periphery and evidence supporting endogenous modulation of pain systems by cannabinoids, provide support that cannabinoids exhibit significant potential as analgesics8-13.

In addition sixteen of 19 randomized controlled trials examining cannabinoids in the treatment of pain have demonstrated a significant analgesic effect , nine of the positive trials involved neuropathic pain 14. Several of these trials examined a cannabinoid extract preparation Sativex15-20 proposed in the current trial.

What is the current standard of care for neuropathic pain caused by chemotherapy?

The current standard of care for neuropathic pain associated with chemotherapy is similar to that for management of chronic neuropathic pain. The approach consists of an interdisciplinary active participatory approach to living with incurable pain. This includes trials of pharmacotherapy (eg. anti-convulsant analgesics, tricyclic antidepressant analgesics and opioids), therapeutic exercise programs and training in coping strategies such as pacing and positive self talk. Such an approach is offered at multidisciplinary pain centres such as the Pain Management Unit (PMU) here at CDHA.

Study question:

Given the limitations of current best practice, the compelling pre-clinical work supporting that cannabinoids exhibit anti-nociceptive effects in neuropathic pain and more specifically in chemotherapy induced neuropathic pain and initial clinical trials supporting that Sativex exhibits efficacy in other types of neuropathic pain we propose a pilot trial of 30 patient to evaluate the effectiveness of Sativex in treatment of neuropathic pain caused by chemotherapy. If there are positive therapeutic effects in the pilot trial, we plan a subsequent randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Neuropathic pain beginning after chemotherapy with paclitaxil, vincristine or cis-platin that has been present for 3 months or longer.
* Presence of allodynia, hyperalgesia or hypoesthesia on sensory testing in the area of pain.
* Moderate to severe pain, as defined by an average 7-day pain score of greater than 4.0 on an 11-point numerical rating scale for pain intensity (NRS-PI).
* Medications must have been stable for at least14 days.
* Ability to follow the protocol
* Willing and able to give written informed consent.

Exclusion Criteria:

* Ischemic heart disease
* Personal history of schizophrenia or psychotic disorder
* Family history of schizophrenia or psychotic disorder in first degree family member (parent, sibling or child)
* Allergy to cannabinoids
* Presence of any other clinically significant medical disorder (other than the cancer requiring chemotherapy) on history or physical exam that would compromise the participants' safety in the trial as judged by the study physician

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2010-06; Primary Completion 2012-12 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Change in the NRS-PI from baseline to the final week of stable dose treatment) | Patients will titrate the dose to a level where they obtain an analgesic effect without limiting side effects (week 3)
Participants gaining a 30% or greater reduction in the NRS-PI | Patients will titrate the dose to a level where they obtain an analgesic effect without limiting side effects (week 3)

SECONDARY OUTCOMES:
Secondary outcome measures will include measures in the remaining domains (suggested by IMMPACT). These include SF36, Quantitative sensory examination, Global Impression of Change, PGIC and Patient Satisfaction Scale, PSS | After stable dosing is achieved (week 3)

CONTACTS AND LOCATIONS:
Overall Officials: Mary E Lynch, MD, Principal Investigator — Nova Scotia Health Authority
Locations (1):
- Queen Elizabeth II Health Sciences Centre, Pain Management Unit, Halifax, Nova Scotia, Canada

REFERENCES:
- [Result] Lynch ME, Cesar-Rittenberg P, Hohmann AG. A double-blind, placebo-controlled, crossover pilot trial with extension using an oral mucosal cannabinoid extract for treatment of chemotherapy-induced neuropathic pain. J Pain Symptom Manage. 2014 Jan;47(1):166-73. doi: 10.1016/j.jpainsymman.2013.02.018. Epub 2013 Jun 4. PMID 23742737